CLINICAL TRIAL: NCT02194855
Title: Effect of Laparoscopic Operation on Rocuronium and Cisatracurium: Pharmacokinetic and Pharmacodynamic Analysis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tingting Wang, Tingting Wang, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TingtingWang
Record Dates: First submitted 2014-07-11; First posted 2014-07-18 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: C.Delivery; Surgery (Previous), Gynecological
Keywords: rocuronium; cisatracurium; pharmacokinetic
MeSH Terms: interventions — Rocuronium; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- laparoscopic operation on rocuronium (Experimental): according different surgical type, all patients were divided into 2 groups: the laparoscopic surgery group and open surgery group.Each group were randomly assigned to the rocuronium group and cisatracurium group.
  Interventions: Drug: rocuronium
- laparoscopic operation on cisatracurium (Experimental): according different surgical type, all patients were divided into 2 groups: the laparoscopic surgery group and open surgery group.Each group were randomly assigned to the rocuronium group and cisatracurium group.
  Interventions: Drug: cisatracurium
- conventional open surgery on rocuronium (Experimental): according different surgical type, all patients were divided into 2 groups: the laparoscopic surgery group and open surgery group.Each group were randomly assigned to the rocuronium group and cisatracurium group.
  Interventions: Drug: rocuronium
- conventional open surgery on cisatracurium (Experimental): according different surgical type, all patients were divided into 2 groups: the laparoscopic surgery group and open surgery group.Each group were randomly assigned to the rocuronium group and cisatracurium group.
  Interventions: Drug: cisatracurium

INTERVENTIONS:
Drug: rocuronium — Rocuronium 0.6 mg.kg-1 was administered within 5 s as an intravenous bolus
  Arms: conventional open surgery on rocuronium; laparoscopic operation on rocuronium
Drug: cisatracurium — cisatracurium 0.15mg.kg-1 was administered within 5 s as an intravenous bolus
  Arms: conventional open surgery on cisatracurium; laparoscopic operation on cisatracurium

SUMMARY:
The investigators investigated whether laparoscopic versus open surgical approaches affected the pharmacokinetic and pharmacodynamic of a single bolus dose of rocuronium or cisatracurium.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology 1-2
* BMI 18-30 kg.m-2
* elective gynaecological operations under general anaesthesia

Exclusion Criteria:

* cirrhosis
* hepatitis
* hepatoma
* heart failure
* arrhythmia
* renal dysfunction
* electrolyte disturbances
* acid-base imbalances
* neuromuscular disorders

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
the blood flow in the right and middle hepatic veins | up to 9 months
  Measurements of the blood flow in the right and middle hepatic veins were performed at baseline and 1,5, 10, 20, 30min after insufflation of carbon dioxide or incise the skin as well as 1 and 5 min after deflation or close the wound.

SECONDARY OUTCOMES:
the plasma Concentration of rocuronium and cisatracurium | up to 9 months
  Venous blood samples (3 ml) were taken 2 min prior to and at 5,30, 60 min following administration of rocuronium/cisatracurium.The aim of the present was to study the blood concentration of rocuronium/cisatracurium in laparoscopic surgery compared with conventional open gynaecological surgery

OTHER OUTCOMES:
pharmacodynamic comparison of rocuronium and cisatracurium | up to 9 months
  This study was undertaken to investigate the duration of action of 0.9 mg.kg-1 rocuronium or cisatracurium 0.15 mg.kg-1 administered during laparoscopic surgery compared with conventional open gynaecological surgery.Adductor pollicis train-of-four responses following ulnar nerve stimulation were monitored with mechanomyography.We recorded the time from the end of injection of rocuronium or cisatracurium to time to recovery of T1, and to recovery to 5% and 25% of baseline height

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, doctor, Principal Investigator — Obstetrics and Gynecology,Fudan University